CLINICAL TRIAL: NCT06893289
Title: The Effect of a Treatment Protocol Focused on Neuromuscular Control Exercises on Pain and Function in a Subgroup of Individuals With Patellofemoral Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Principal Investigator, Ana Luiza Costa e Silva Cabral, PhD candidate, Universidade do Porto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023.00945.BD
Record Dates: First submitted 2025-03-10; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Patellofemoral Pain
Keywords: Patellofemoral pain; Electromyography; Kinematics; Kinetics; Neuromuscular control; PFP subgroups
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients will be blinded to group allocation, ensuring that they will not know which exercises will be performed by the other group, and thus the interventions will be administered separately to members of each treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neuromuscular control exercises (Experimental)
  Interventions: Other: Exercise
- Muscle strengthening (Active Comparator)
  Interventions: Other: Muscle strengthening

INTERVENTIONS:
Other: Exercise — Balance and proprioceptive exercises
  Arms: Neuromuscular control exercises
Other: Muscle strengthening — Strengthening of the lower limb muscles
  Arms: Muscle strengthening

SUMMARY:
Patellofemoral Pain (PFP) is one of the most common causes of knee pain and is significantly present in recreational athletes who have previously been categorized as being in a subgroup of PFP. Understanding which intervention is most appropriate for this subgroup could give us important information about subgroup-based treatments, which are not yet described in the literature. Therefore, the aim of this study is to analyze the effect of two exercise interventions in a PFP subgroup: one focusing on neuromuscular control exercises and the other focusing on muscle strengthening.This study will recruit 10 individuals to each exercise group, and will assess pain, function, muscle activity and joint kinematics pre and post intervention. Mixed Model ANOVA tests will be used to determine the responses to the two interventions between the two groups over a 6-week treatment time.

DETAILED DESCRIPTION:
This study proposes a treatment protocol focused on neuromuscular control in a subgroup of individuals with PFP and may provide important information on the effectiveness of different treatment approaches for patellofemoral pain. It would be interesting to establish objectives according to clinical findings, and thus identify the best treatment protocols for specific subgroups of PFP. For a long time, the focus of rehabilitation has been on decreasing knee pain and strengthening the muscles around the knee to improve knee joint function (Piva et al., 2009) in a generalized way for all individuals with PFP. However, with recent information in the literature on the presence of subgroups, a study with a treatment protocol focused on neuromuscular control directed at a subgroup has not yet been carried out, which is the objective of this work. Thus, the hypothesis to be tested is that individuals from a PFP subgroup will present better results with neuromuscular control exercises than those performing muscle strengthening in the same treatment period.

The aim of this study is to compare the effects of two 6-week treatment protocols a) based on neuromuscular control exercises, and b) muscle strengthening on outcome measures of pain, function and biomechanical variables in a subgroup of individuals with PFP during stair ascent and descent.

-Detailed Description This study will be carried out at the Porto Biomechanics Laboratory (LABIOMEP) and at the gym of the Faculty of Sports (FADEUP) of University of Porto. The recruitment of volunteers for this project will take place in the city of Porto, Portugal. Participants will be invited to participate in the study if they self-report anterior knee pain exacerbated during a squatting test and/or during any sporting practice. Folders with all the information necessary for recruitment will be distributed among the academic and general community, recreational athletes during sporting events and on social media.

Sample calculation A sample size calculation was performed based on the minimal detectable change on the Visual Analog Pain Scale (VAS). Data from a previous study indicate that the mean VAS score in patients with PFP was 4.3 ± 1 cm (Crossley et al. 2004), with 30% of the maximum score of the VAS-pain considered to be the detectable change. The sample size for each group to achieve a 90% power at the 0.05 level of significance was determined to be 8 patients. Thus, the sample will consist of 20 volunteers (ten per group) of both sexes diagnosed with PFP.

Inclusion criteria Men and women aged 18-40 years old that can give informed written consent. Clinical diagnosis of unilateral or bilateral PFP longer than 3 months (exemplified in the following sections).

Anterior or retropatellar pain reported on at least two of the following activities: prolonged sitting, ascending or descending stairs, running, kneeling and hopping/jumping.

At least two of the three following clinical examination findings:

* Pain during resisted isometric quadriceps contraction
* Pain with palpation of the posterior borders of the patella
* Pain during squatting Classified as a subgroup of PFP (exemplified in the following sections).

Exclusion criteria Individuals who are not part of a PFP group Previous knee surgery and participants awaiting surgery for another lower limb joint problem Ligamentous instability and/or internal pathology History of patella subluxation or dislocation Joint effusion when the midpatellar girth is 5% or more than the non-involved knee True knee joint locking and/or giving way Coexistent acute illness or chronic disease Bursitis, patella or iliotibial tract tendinopathy, Osgood-Schlatter's disease, Sinding-Larsen-Johansson Syndrome, muscle tears or symptomatic knee plicae Pregnancy or breast feeding

Clinical diagnosis of PFP The specific diagnosis of PFP will be made according to the recommendations of the Clinical Practice Guideline of Patellofemoral Pain (Willy et al. 2019).

1. the presence of retropatellar or peripatellar pain,
2. reproduction of retropatellar or peripatellar pain with squatting, stair climbing, prolonged sitting, or other functional activities loading the patellofemoral joint in a flexed position, and
3. exclusion of all other conditions that may cause anterior knee pain, including tibiofemoral pathologies.

Also, the patellar tilt test will be used to verify mobility of the patella to support the diagnoses.

Clinical classification of a subgroup of PFP The classification into subgroups will be performed using the six clinical tests described by Selfe et al. 2016. The therapist manual of the Target Intervention for Patellofemoral Pain Syndrome (TIPPS) was made available by the authors of the original study and will be used as a guide to stratify individuals with PFP.

The first day of pre-intervention assessments will be carried out at the gym of the Faculty of Sports (FADEUP) of University of Porto. A physical therapist will access sociodemographic, anthropometric and contact data from each patient through an evaluation form. In no field of the evaluation form will the participant be identified. Baseline data will be collected following the recommendations of the REPORT-PFP checklist of items recommended for quantitative studies with individuals with PFP (Barton et al. 2021). The instruments that will be used to collect baseline symptoms are described in the following table. The administration method of all instruments that will be used to assess baseline symptoms is self-reportable.

Then, eligibility criteria, clinical diagnosis of PFP, and classification of subgroup according to the previous sections will be verified. The affected/most affected limb will be evaluated. All data from the first day of assessment will be analyzed and the individual will be invited to the second day of assessment only if they meet the eligibility criteria. If the individual is interested in participating, they will be asked to sign the informed consent form on the second day of pre-intervention assessment.

The second day of pre-intervention assessment will be carried out at the Porto Biomechanics Laboratory (LABIOMEP) of the University of Porto. The individual will sign the informed consent form and will then be prepared for the collection of kinetic and kinematic data. These data will be collected during stair ascent-descent.

Kinematic data will be recorded using a 3D motion capture system (three Oqus 310+ and nine Oqus 400 Qualisys infrared cameras, AB, Gothenburg, Sweden), sampling at 100 Hz. Thus, to obtain a three-dimensional (3D) biomechanical model, the 3D trajectories of passive retro-reflective markers will be captured. For the placement of the markers, the Calibrated Anatomical System Technique that allow for segmental kinematics to be tracked in 6-degrees of freedom will be used. It will be positioned on the anterior superior iliac spine, posterior superior iliac spine, greater trochanter, medial and lateral femoral epicondyles, medial and lateral malleoli, the medial aspect of the head of the 1st metatarsal, the lateral aspect of the head of the 5th metatarsal, the dorsum of the foot and the calcaneus. Additionally, clusters of four noncollinear markers will be attached to each of the body segments (Richards et al. 2018).

For kinetic data, a four-step staircase with a force platform embedded on each step will be used (two Bertec, OH, USA and two AMTI, MA, USA) sampling at 2000 Hz. The steps have a riser height of 17 cm, run of 25 cm, and width of 60 cm.

Electromyography evaluation will be made with four dEMG Delsys Trigno Wireless sensors positioned over the Vastus Medialis (VM) and Vastus Lateralis (VL) muscles of both limbs. The positioning of the electrodes will be carried out according to SENIAM - Surface Electromyography for the Non-Invasive Assessment of muscles (Hermens et al., 2000).

In the revaluation, the baseline symptoms (pain, function, kinesiophobia, IPAQ, GROC), biomechanical and electromyography assessments will be performed again.

Randomization The stratified randomization method will be performed to balance the two treatment groups according to gender (Kang, Ragan, e Park 2008). Randomization will be performed after baseline and biomechanical assessments, and patients will be blinded to group allocation, ensuring that they will not know which exercises will be performed by the other group, and thus the interventions will be administered separately to members of each treatment group (Baldon et al. 2014).

Treatment protocols The individuals will be separated into two groups: group 1 (G1) - usual treatment group; and group 2 (G2) - neuromuscular control exercise group. Both groups will undergo 6 weeks of treatment, with 3 sessions of 60 minutes per week (Yosmaoğlu et al. 2019). In each session, 10 minutes of warm-up will be performed before the start of the intervention.

During the study period, volunteers will be asked not to seek another type of treatment for knee pain and to maintain their regular daily activities. Each volunteer will be supervised by a researcher trained specifically for the treatment under study. The Template for Intervention Description and Replication (TIDieR) will be used to describe the interventions (Hoffmann et al. 2014). If patients report severe pain at any point, the intensity of the exercise will be reduced so that they can perform the movement without pain.

Intended statistical analysis Descriptive statistics of means and standard deviations will be obtained for each outcome measure. Shapiro-Wilk tests will be used to screen the data for normality. Differences in biomechanical and knee pain parameters will be examined using 2 (pre-post intervention) x2 (subgroup) Mixed Model ANOVA tests. Statistical significance will be accepted at the P≤0.05 level. Effect sizes will be calculated using partial Eta2 (pη2). Effect sizes will be contextualized using the following guidelines: small = 0.01, medium = 0.06 and large = 0.14 (Cohen, 1988). All statistical analysis will be performed using SPSS v24.0 (SPSS Inc, Chicago, USA).

ELIGIBILITY:
Inclusion Criteria Men and women aged 18-40 years old that can give informed written consent. Clinical diagnosis of unilateral or bilateral PFP longer than 3 months (exemplified in the following sections).

Anterior or retropatellar pain reported on at least two of the following activities: prolonged sitting, ascending or descending stairs, running, kneeling and hopping/jumping.

At least two of the three following clinical examination findings:

* Pain during resisted isometric quadriceps contraction
* Pain with palpation of the posterior borders of the patella
* Pain during squatting Classified as a subgroup of PFP.

Exclusion Criteria Individuals who are not part of a PFP group Previous knee surgery and participants awaiting surgery for another lower limb joint problems Ligamentous instability and/or internal pathology History of patella subluxation or dislocation Joint effusion when the midpatellar girth is 5% or more than the non-involved knee True knee joint locking and/or giving way Coexistent acute illness or chronic disease Bursitis, patella or iliotibial tract tendinopathy, Osgood-Schlatter's disease, Sinding-Larsen-Johansson Syndrome, muscle tears or symptomatic knee plicae Pregnancy or breast feeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Pain at rest | From enrollment to the end of treatment at 6 weeks
  Numerical Pain Rating Scale (NPRS)
Pain during activity | From enrollment to the end of treatment at 6 weeks
  Numerical Pain Rating Scale (NPRS)
Function | From enrollment to the end of treatment at 6 weeks
  Knee injury and Osteoarthritis Outcome Score - KOOS

SECONDARY OUTCOMES:
Kinematic data - hip, knee and ankle angles | From enrollment to the end of treatment at 6 weeks
  Motion capture system
Kinetic data - hip, knee, and ankle moments and ground reaction forces | From enrollment to the end of treatment at 6 weeks
  Force platforms
Muscular activity | From enrollment to the end of treatment at 6 weeks
  Electromyography system

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Sport of University of Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No